CLINICAL TRIAL: NCT00669357
Title: AbioCor Implantable Replacement Heart
Status: No longer available | Type: Expanded Access
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: H040006
Record Dates: First submitted 2008-04-25; First posted 2008-04-30 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Severe Biventricular End Stage Heart Disease
Keywords: End stage heart disease

INTERVENTIONS:
Device: Abiocor Implantable Replacement Heart — Replacement of heart

SUMMARY:
Abiocor is a post market approval study for an Implantable Replacement Heart. This post approval study is currently on hold.

ELIGIBILITY:
Inclusion Criteria:

* Patients in severe biventricular end stage heart disease who are not cardiac transplant candidates and who are adults less than 75 years old, require multiple inotropic support, are not treatable by LVAD destination therapy, and are not weanable from biventricular support if on such support.

Exclusion Criteria:

* Patients with other irreversible end organ dysfunctions that would compromise survival, having in clinical assessment a more than 30% chance of survival beyond 30 days, inadequate psychosocial support, or patients in whom fit is a problem, based on preoperative noninvasive anatomical assessment showing that the thoracic volume is unable to accommodate the device.

Max Age: 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult